CLINICAL TRIAL: NCT00225472
Title: Organ Preservation Media Investigation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 2002-566
Record Dates: First submitted 2005-09-13; First posted 2005-09-23 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Kidney Transplant

INTERVENTIONS:
Device: Modified Viaspan

SUMMARY:
Kidney transplantation remains limited by four problems: 1) a too high rate of delayed graft function, 2) early loss of kidneys from chronic rejection, 3) donor kidney shortages, and 4) the need for immunomodulating treatments. Improved cold storage methods can significantly impact on the first 3 of these 4 major problems. The device to be tested is a modification of the existing Viaspan organ preservation solution. The modification of this solution combines four compounds: Bovine neutrophil peptide-1 (BNP-1), Substance P (SP), Insulin-like growth factor-1 (IGF-1), and Nerve Growth Factor (NGF). This solution will be added to Viaspan for preservation of donor kidneys. Preclinical data indicates that trophic factor deprivation during cold storage is a significant and previously unrecognized mechanism of injury in cold stored kidneys. The aim of this study is improved graft function, decreasing early graft loss due to rejection, and decreasing the donor organ shortage.

ELIGIBILITY:
Inclusion Criteria:

* first renal transplant, PRA's <20%

Exclusion Criteria:

* PRA's greater than 20%
* Subjects who are receiving a non-primary renal transplant
* Subjects under the age of 18
* Pregnant or nursing women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2004-06; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Dalessandro, MD, Principal Investigator — University of Wisconsin Medical School
Locations (1):
- University of Wisconsin Hospital and Clinics, Madison, Wisconsin, United States